CLINICAL TRIAL: NCT02819609
Title: Comparing Patient-Centered Outcomes After Treatment for Uterine Fibroids
Status: Completed | Type: Observational
Sponsor: Quintiles, Inc. (Industry)
Collaborators: Center for Medical Technology Policy (Unknown); Duke University (Other)
Responsible Party: Principal Investigator, Priscilla Velentgas, Senior Director of Epidemiology and Health Outcomes, Quintiles, Inc.
Other Study IDs: CE-12-11-4430
Record Dates: First submitted 2016-02-12; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — Uterine Myomectomy; Endometrial Ablation Techniques; Uterine Artery Embolization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- Myomectomy: Women with uterine fibroids who underwent myomectomy as their index procedure as part of their routine clinical care
  Interventions: Procedure: myomectomy
- Endometrial ablation: Women with uterine fibroids who underwent endometrial ablation as their index procedure as part of their routine clinical care
  Interventions: Procedure: endometrial ablation
- Uterine artery embolization: Women with uterine fibroids who underwent uterine artery embolization as their index procedure as part of their routine clinical care
  Interventions: Procedure: uterine artery embolization
- MRI-guided focused ultrasound ablation: Women with uterine fibroids who underwent MRI-guided focused ultrasound ablation as their index procedure as part of their routine clinical care
  Interventions: Procedure: MRI-guided focused ultrasound ablation

INTERVENTIONS:
Procedure: myomectomy — Myomectomy as part of routine clinical care
  Groups: Myomectomy
Procedure: endometrial ablation — Endometrial ablation as part of routine clinical care
  Groups: Endometrial ablation
Procedure: uterine artery embolization — Uterine artery embolization as part of routine clinical care
  Groups: Uterine artery embolization
Procedure: MRI-guided focused ultrasound ablation — MRI-guided focused ultrasound ablation as part of routine clinical care
  Groups: MRI-guided focused ultrasound ablation

SUMMARY:
The purpose of this observational, retrospective database study of patients with uterine fibroids is to compare the durability of symptom relief after uterus-conserving treatments for symptomatic fibroids in terms of incidence of, and time to, new or recurrent symptoms and subsequent procedures and evaluate the effect stakeholder participation had on the research process.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with a diagnosis of uterine fibroids at any time and at least 1 office visit during study time period
* At least 1 of the procedures of interest occurring between January 1, 2005 - December 31, 2011
* ≥ 18 years and < 55 years of age at the index date

Exclusion Criteria:

* Patients with a diagnosis of gynecologic cancer (ovarian, uterine, cervical)
* First recorded diagnosis of uterine fibroids occurring beyond four weeks after the Index Date ONLY for patients who underwent endometrial ablation or hysterectomy
* Patients with a record of any procedures of interest occurring before January 1, 2005

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The patient population for the retrospective data analysis was uterine fibroid patients who have a record of at least 1 of the procedures of interest occurring during the time period of January 1, 2005 - December 31, 2011, with the first instance being designated as the index date. The study time period spanned from January 1, 2004 - December 31, 2013 to allow for 12 months pre-index for evaluating baseline demographic and clinical characteristics and 24 months post-index, ensuring a minimum of 2 years follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 12234 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of uterine fibroids patients who experience new or recurrent symptoms after uterus-conserving treatments (myomectomy, endometrial ablation, uterine artery embolization, magnetic resonance imaging [MRI]-guided focused ultrasound ablation) | Minimum of two years after index procedure
Time to new or recurrent symptoms after uterus-conserving treatments (myomectomy, endometrial ablation, uterine artery embolization, magnetic resonance imaging [MRI]-guided focused ultrasound ablation) | Minimum of two years after index procedure
Number of uterine fibroids patients who experience a subsequent procedure after uterus-conserving treatments (myomectomy, endometrial ablation, uterine artery embolization, magnetic resonance imaging [MRI]-guided focused ultrasound ablation) | Minimum of two years after index procedure
Time to a subsequent procedure after uterus-conserving treatments (myomectomy, endometrial ablation, uterine artery embolization, magnetic resonance imaging [MRI]-guided focused ultrasound ablation) | Minimum of two years
Effect of stakeholder participation in the research process | From first stakeholder conference (April 2014) to final stakeholder conference (November 2015)